CLINICAL TRIAL: NCT00786708
Title: Sensitivity and Specificity of Neutrophil Gelatinase-Associated Lipocalin (NGAL) in an Emergency Room Population
Brief Title: Sensitivity and Specificity of NGAL in an Emergency Room Population
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Abbott (Industry); Charite University, Berlin, Germany (Other); Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Nickolas, Assistant Professor of Medicine, Department of Medicine, Nephrology, Columbia University
Other Study IDs: AAAC1584
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Azotemia; Renal Insufficiency, Chronic; Renal Failure, Acute; Hydronephrosis
Keywords: renal; kidney; lipocalin; urine; biomarker; Azotemia; Renal insufficiency, chronic; Renal failure, acute; Hydronephrosis
MeSH Terms: conditions — Azotemia; Renal Insufficiency, Chronic; Acute Kidney Injury; Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NGAL: Urine that would otherwise be discarded will be obtained from a convenience sample of patients admitted to the hospital through the emergency room who meet the inclusion / exclusion criteria for this study.

SUMMARY:
Hypothesis: In patients that present to an urban emergency room, a single urine neutrophil gelatinase-associated lipocalin (NGAL) measurement can classify their kidney disease as stable chronic kidney disease, acute tubular necrosis, urinary outlet obstruction or pre-renal azotemia.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether urinary NGAL levels are able to distinguish the classical categories of renal disease. Previous studies have strongly suggested that this protein marks those with fulminant renal dysfunction with greater sensitivity and time resolution than currently used markers. Studies to date have been in highly selected populations: children and adults following cardiac surgery, infants with cardiovascular anomalies, and patients with known chronic kidney disease. Demonstration of similarly robust sensitivity and specificity in a broad Emergency Room population would strengthen the conception of NGAL as a marker of early or advancing kidney dysfunction. Most importantly, if NGAL can distinguish between types of renal disease at presentation in the ER, it might have important implications regarding ER management of these common presentations. For example, it could reduce diagnostic ambiguity and lag time from hours or days to seconds.

ELIGIBILITY:
Inclusion Criteria:

A. Must be greater than or equal to 18 years of age

B. Must satisfy the following age and sex stratified serum creatinine levels:

1. men between ages 18 and 50 with serum creatinine greater than 1.2mg/dl
2. women between ages 18 and 50 with serum creatinine greater than 1.2mg/dl
3. men older than 50 with serum creatinine greater than 1.0mg/dl
4. women older than 50 with serum creatinine greater than 0.8mg/dl

C. All pts greater than or equal to 18 years of age without kidney failure defined by B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital through the emergency room who meet the inclusion / exclusion criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 2304 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The correlation of elevated urine NGAL with the diagnosis of intrinsic acute kidney injury. | Assessed retrospectively after patient is discharged

SECONDARY OUTCOMES:
The correlation of urine NGAL and inpatient morbidity assessed by nephrology consultation and other factors such as dialysis initiation and intensive care unit stay. | Assessed retrospectively after patient is discharged

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Nickolas, MD, MS, Principal Investigator — Columbia University; Jonathan Barasch, MD, PhD, Principal Investigator — Columbia University
Locations (3):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
- Charite University Medical Center, Berlin, Germany

REFERENCES:
- [Result] Nickolas TL, Schmidt-Ott KM, Canetta P, Forster C, Singer E, Sise M, Elger A, Maarouf O, Sola-Del Valle DA, O'Rourke M, Sherman E, Lee P, Geara A, Imus P, Guddati A, Polland A, Rahman W, Elitok S, Malik N, Giglio J, El-Sayegh S, Devarajan P, Hebbar S, Saggi SJ, Hahn B, Kettritz R, Luft FC, Barasch J. Diagnostic and prognostic stratification in the emergency department using urinary biomarkers of nephron damage: a multicenter prospective cohort study. J Am Coll Cardiol. 2012 Jan 17;59(3):246-55. doi: 10.1016/j.jacc.2011.10.854. PMID 22240130